CLINICAL TRIAL: NCT01333800
Title: Phase 4 Cost-effectiveness Study of Beclomethasone Versus Ciclesonide as Controller Medications in Pediatric Asthma in a Hospital in Bogotá
Brief Title: Cost-effectiveness Study of Beclomethasone Versus Ciclesonide as Controller Medications in Pediatric Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grünenthal Colombiana S.A. (Industry)
Responsible Party: Francisco Hinestrosa, Grünenthal Colombiana S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO-AL-FE-001
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; ciclesonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciclesonide (Active Comparator)
  Interventions: Drug: Ciclesonide
- Beclomethasone (Placebo Comparator)
  Interventions: Drug: Beclomethasone

INTERVENTIONS:
Drug: Beclomethasone — 200 to 400 mcg per day for 6 months
  Arms: Beclomethasone
Drug: Ciclesonide — 80 to 160 mcg per day for 6 months
  Arms: Ciclesonide

SUMMARY:
The Objective was to Develop a Cost-Effectiveness study that compares Ciclesonide and Beclomethasone in pediatric asthma control.

DETAILED DESCRIPTION:
Cost-effectiveness study, of cohorts, observational, analytic, prospective, from health institution perspective. Based on published data related to percentage of patients free of crisis for both molecules, it was estimated that the sample size to detect significant differences between the two alternatives was 20 patients per alternative. Medical records of 94 patients with diagnosis of uncontrolled asthma were included, aged between 6 and 15 years, 47 received Beclomethasone randomly, and 47 received Ciclesonide randomly, treatment physician was blind related to this assignation, both cohorts were followed for 6 months, and primary effectiveness variable was defined as number of patients free of crisis with each alternative. Cost generating variables were defined as medication use, and hospital stay. Decision analysis was based on a decision tree.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled asthma diagnosis
* Patients with only one controller medication

Exclusion Criteria:

* Patients without lung infection
* Patients without antibiotic use

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness measured as number of patients free of asthmatic crisis with each molecule during the study period | 6 months
  Effectiveness was assesed counting number of patients that were free of asthmatic crisis for each steroid ciclesonide and beclomethasone during 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Hinestrosa, MD,MSc, Principal Investigator — Grünenthal Colombiana S.A.
Locations (1):
- Hospital San Rafael, Bogotá, Colombia